CLINICAL TRIAL: NCT05903391
Title: Splint Users' Satisfaction and Functional Status With Custom Finger Splints: A Feasibility and Comparison Study
Brief Title: Splint Users' Satisfaction and Functional Status With Custom Finger Splints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Natasha Irani, OTD, OTR/L: Occupational Therapist, Endeavor Health
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: EH23-047
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Hypermobility of Interphalangeal Joints; Swan-Neck Deformity
Keywords: 3d-printing; technology; finger splints; hypermobile joints

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 3D-Printed Finger Splints (Experimental): Participants who wear the experimental customizable 3D-printed finger splints
  Interventions: Device: 3D-Printed Finger Splints
- Conventional Finger Splints (Active Comparator): Participants who wear the control, conventionally made finger splints
  Interventions: Device: Conventional Finger Splints

INTERVENTIONS:
Device: 3D-Printed Finger Splints — The intervention is wearing a novel finger splint produced by a 3D-printer
  Arms: 3D-Printed Finger Splints
Device: Conventional Finger Splints — This intervention is wearing a finger splint produced by a conventional method using thermoplastic material typically used in a clinical setting
  Arms: Conventional Finger Splints

SUMMARY:
This feasibility and non-randomized comparison study explores the possible benefits of splint design and production by 3D-printing in a clinical setting and looks at splint users' experiences with customizable 3D-printed finger splints compared to conventionally made splints. Fifty participants with a hyperextended finger condition are assigned by researcher to either an interventional group (customizable 3D-printed finger splint) or a control group (conventional thermoplastic finger splint). Participants will wear assigned splint for 1 month. Functional status and satisfaction with splint will be assessed at the end of the 1-month duration in the form of surveys on satisfaction and functional status participants will be asked to complete. The findings will contribute to evidence that customizable 3D-printed finger splints can serve as a feasible, cost-effective option to improve patient satisfaction and functional status. It will further justify the need for the application of 3D-printing in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* 18 years or older
* Finger proximal interphalangeal joint (PIP) joint hyperextension (with or without swan-neck deformity)
* Pregnant or not pregnant women
* Able to tolerate a finger orthosis over the course of 1 month
* Not decisionally impaired
* Have or have not previously worn a finger orthosis for symptoms

Exclusion Criteria:

* Non-fluent in English
* Decisionally impaired
* Younger than 18 years old
* No proximal interphalangeal joint (PIP) joint finger hyperextension
* Unable to tolerate a finger orthosis over the course of 1 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Modified Version of Orthotics and Prosthetics User Survey - Satisfaction with Device | 1 month
  A modified version of a Self-report questionnaire which measures participants satisfaction with assigned splint device
Modified Version of Orthotics and Prosthetics User Survey - Functional Status | 1 month
  A modified version of a Self-report questionnaire which measures participants' functional status during the duration of time wearing assigned finger splint device

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Swedish Hospital Part of NorthShore University HealthSystems, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois

IPD SHARING:
Plan to Share IPD: No